CLINICAL TRIAL: NCT04446234
Title: Atypical Antipsychotics Influence on the Safety of the Heart and Monitoring Indicators Model Building
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YG2019QNB07
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-06

CONDITIONS: Schizophrenia
Keywords: Atypical antipsychotics; Cardiac safety; Model building
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Aripiprazole; ziprasidone; Amisulpride; Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Risperidone (Experimental): Risperidone tablet
  Interventions: Drug: Risperidone
- Aripiprazole (Experimental): Aripiprazole tablet
  Interventions: Drug: Aripiprazole
- Ziprasidone (Experimental): Ziprasidone tablet
  Interventions: Drug: Ziprasidone
- Amisulpride (Experimental): Amisulpride tablet
  Interventions: Drug: Amisulpride
- Quetiapine (Experimental): Quetiapine tablet
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Risperidone — Use medicine according to patients condition
  Arms: Risperidone
Drug: Aripiprazole — Use medicine according to patients condition
  Arms: Aripiprazole
Drug: Ziprasidone — Use medicine according to patients condition
  Arms: Ziprasidone
Drug: Amisulpride — Use medicine according to patients condition
  Arms: Amisulpride
Drug: Quetiapine — Use medicine according to patients condition
  Arms: Quetiapine

SUMMARY:
The purpose of this study was to investigate the effect of atypical antipsychotics on cardiac safety. The secondary purpose was to understand the rate of QTc prolongation in electrocardiogram induced by atypical antipsychotics. And try to construct the model of cardiac monitoring index. We conducted a randomized trial in which patients with schizophrenia who were first on or off medication for more than two weeks took a single atypical antipsychotic (Risperidone, Aripiprazole, Ziprasidone, Amisulpride, Quetiapine) for 12 weeks and monitored changes in biochemical, electrocardiogram and other indicators. And then 50 patients with adverse cardiac reactions (ADRs) taking antipsychotics were selected to review the data, analyze and construct a monitoring model.

We hypothesized that atypical antipsychotics with different mechanisms of action have different effects on cardiac safety in patients with schizophrenia, and that they are applicable to different populations. The monitoring index model can reduce the occurrence of cardiotoxicity and improve the prognosis.

DETAILED DESCRIPTION:
Atypical antipsychotics, also known as new antipsychotics, are a group of drugs that act on the central nervous system to treat schizophrenia, psychotic disorder or bipolar disorder. Compared with typical antipsychotics, atypical antipsychotics have the advantages of good efficacy and fewer side effects. Therefore, currently, atypical antipsychotics are widely used in clinical practice. In recent years, the effects of atypical antipsychotics on metabolism and cardiovascular system have attracted more and more clinical attention. Studies have found that long-term use of atypical antipsychotics can lead to arrhythmias, drug-induced myocarditis, and even cardiac arrest. Since antipsychotics can cause cardiac adverse events in patients with schizophrenia, accompanied by medical complications, resulting in a generally shorter life span of 15-25 years compared with the general population, cardiac safety assessment of drugs for patients with schizophrenia is becoming increasingly important. But the domestic study of antipsychotics in the cardiovascular field, especially about the safety of heart systemic evaluation are few and far between, so this research has focused on patients with schizophrenia in China people use different mechanisms of atypical antipsychotics (Risperidone, Aripiprazole, Ziprasidone, Amisulpride, Quetiapine) on heart safety.

In the first stage, a total of 350 schizophrenia patients were enrolled who were either not on medication for the first time or stopped for more than 2 weeks. They were treated with atypical antipsychotics respectively, follow-up of 12 weeks, evaluating the effects of antipsychotics on cardiac function and structure in patients with schizophrenia from general data, biochemistry, electrocardiogram, etc. In the second stage, 50 patients of adverse cardiac reactions caused by taking antipsychotics were selected from enrolled subjects, and a retrospective analysis(day1, week4, week12, and week24) was conducted to try to build a cardiac safety detection indicator model, so as to understand the impact of antipsychotics on cardiac safety. More rational use of antipsychotics in the context of ensuring clinical efficacy and minimum side effects, and the use of monitoring indicator models to reduce the occurrence of cardiac toxicity, improve the safety of antipsychotics in use.

ELIGIBILITY:
Inclusion Criteria:

* Phase one:Effects of different types of atypical antipsychotics on cardiac safety.

  1. Meet the diagnostic of "schizophrenia" according to DSM-IV and fail to take medication in the first episode or stop taking medication for more than 2 weeks
  2. Han ethnic, 18-45 years old;
  3. Exclude persons with mental disorders caused by organic diseases, drugs or alcohol, and other mental disorders, and serious suicide attempts.
  4. Willing to participate in the trial and receive treatment;
  5. Course of disease within 2 years;
  6. Able to communicate effectively with the researcher and complete the written informed consent signed by hand.

Phase two:Construction of cardiac safety monitoring model

1. Meet the diagnostic of "schizophrenia" according to DSM-IV and fail to take medication in the first episode or stop taking medication for more than 2 weeks
2. Han ethnic, 18-45 years old;
3. Exclude persons with mental disorders caused by organic diseases, drugs or alcohol, and other mental disorders, and serious suicide attempts.
4. Willing to participate in the trial and receive treatment;
5. Serious arrhythmia, myocarditis, cardiomyopathy and cardiac insufficiency during taking medicine;
6. Able to communicate effectively with the researcher and complete the written informed consent signed by hand.

Exclusion Criteria:

* (1) Participating in other clinical studies; (2) Combination of DSM-IV diagnoses other than schizophrenia; (3) History of heart disease; (4) History of drug abuse in the previous 6 months; (5) Pregnant or in the first three months of lactation; (6) Combination of antipsychotics, mood stabilizers and antidepressants was used in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac QTc(corrected QT interval) interphase changes after drug administration. | baseline, week2,4, 8, 12，24
  Cardiac QTc interphase changes during the study duration

SECONDARY OUTCOMES:
Biochemical index： BNP(Brain Natriuretic Peptide) | baseline, week2,4, 8, 12，24
  Changes of biochemical indexes during the study duration
Biochemical index：troponin | baseline, week2,4, 8, 12，24
  Changes of biochemical indexes during the study duration
Biochemical index： myoglobin | baseline, week2,4, 8, 12，24
  Changes of biochemical indexes during the study duration
Electrocardiogram：Heart rate | baseline, week2,4, 8, 12，24
  Changes of ECG indicators during the study duration
Echocardiographic: EF(Ejection Fraction) value | baseline, week2,4, 8, 12，24
  Changes of cardiac ultrasound indicators during the study duration

CONTACTS AND LOCATIONS:
Overall Officials: LV QINYU, Principal Investigator — SHANGHAI MENTAL HEALTH CENTRE
Locations (1):
- CHINA, Shanghai, Minhang, China